CLINICAL TRIAL: NCT00443066
Title: Clinical Study of Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: The Spinal Muscular Atrophy Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AAAB1635; CU52029001 (Other: SMA)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Spinal Muscular Atrophy
Keywords: pediatric; neuromuscular disease
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and skin tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to prepare for clinical trials where SMA patients are asked to join the research effort. The visits will include questions, physical exam, blood drawing, and sometimes X-rays and a skin biopsy. The investigators will use modern computer methods to process the information during which the investigators will plan a clinical trial. Once the clinical trial begins, the investigators will offer SMA patients participation if they meet the criteria for that trial.

Identifying an effective SMA treatment is very important because there is currently none. Clinical trials are the only way to decide whether a new treatment works in SMA patients or not.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is one of the most devastating neurological diseases of childhood. Affected infants and children suffer from progressive muscle weakness caused by degeneration of lower motor neurons in the spinal cord and brainstem. Clinically, four phenotypes are distinguished within the continuous spectrum of disease severity based on the age of onset and the highest motor milestone ever achieved. SMA is caused by homozygous deletion of the survival motor neuron-1 (SMN1) gene. A related gene, SMN2, produces low levels of full-length SMN protein due to inefficient splicing. There is an inverse correlation between SMN copy number and disease severity, presumably mediated by levels of full length SMN protein. Therefore, increasing the amount of full-length SMN protein is a promising treatment strategy. Several drugs targeting splicing efficiency have resulted in increased SMN protein in preclinical assays and are now awaiting clinical testing.

With the future objective to conduct clinical trials in SMA, the proposed project has 3 specific aims: 1) To establish a web-based database that will serve to enroll the patient population and that will facilitate timely recruitment for future clinical trials; (2) to plan for clinical trials by a) developing reliable outcome measures, and (b) establishing the infrastructure needed to carry out efficient clinical trials, (c) convening meetings of preclinical and clinical researchers involved in SMA drug development to select candidate drugs, and (3) to characterize the patient population from a clinical and molecular point of view.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of Spinal Muscular Atrophy
* Genetic diagnosis of SMN gene deletion
* Parents or if applicable subjects must give informed consent
* must be capable of complying with the study procedures
* Female subjects of child-bearing potential must agree to undergo pregnancy test prior to radiological studies
* Diagnosis of SMA before age 19 years

Exclusion Criteria:

* Unstable medical condition precluding participation
* Significant respiratory compromise that would interfere with safe travel to site of evaluation. (The clinical site PI decides when air travel is not recommended and when the patient's location is not within a reasonably safe driving distance (upper limit 150-250 miles)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People diagnosed with Spinal Muscular Atrophy types I, II, or III before the age of 17.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2005-05; Primary Completion 2011-08-17 (Actual); Study Completion 2011-08-17 (Actual)

PRIMARY OUTCOMES:
Hammersmith Functional Motor Scale Expanded (HFMSE) | Up to 36 months
  For SMAII/III patients over 2 years of age, we will additionally administer the Hammersmith SMA functional motor scale (H-SMA-FMS), a disease-specific instrument.
Gross Motor Function Scale (GMFM) | Up to 36 months
  The GMFM contains 88 items in 5 dimensions: (A) lying and rolling, (B) sitting, (C) crawling, (D) standing, and (E) walking.

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C De Vivo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University SMA Clinical Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No